CLINICAL TRIAL: NCT04052113
Title: Real World Evidence of PD-L1, TMB Prevalence and Efficacy of 1st Line Chemotherapy in These High or Low Population for Stage IV Urothelial Cancer
Acronym: YODO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D419BR00014
Record Dates: First submitted 2019-07-22; First posted 2019-08-09 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Urologic Neoplasms
Keywords: Real world, PD-L1, TMB, Stage IV, urothelial cancer, Japanese
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No

SUMMARY:
This study is a multi-center, non-interventional study. Patients' background, treatment pattern, treatment outcome, efficacy will be collected from medical records in Stage IV urotherial (UC) patients. Archived patient's formalin-fixed paraffin-embedded (FFPE) primary tumor samples will be collected to assay PD-L1 expression and next generation sequencer (NGS) assay for tumor mutation burden (TMB).

DETAILED DESCRIPTION:
This study is a multi-center, non-interventional study. Patients' background, treatment pattern, treatment outcome, efficacy will be collected from medical records in Stage IV urotherial (UC) patients. Archived patient's formalin-fixed paraffin-embedded (FFPE) primary tumor samples will be collected from each site and conduct programmed cell death 1 ligand 1 (PD-L1) assay and next generation sequencer (NGS) assay for tumor mutation burden (TMB). Based on these data, prevalence of PD-L1, TMB and overall survival (OS), progression free survival (PFS) from start of 1st line treatment in stage IV will be assessed.

In this study, 150 patients will be enrolled from approximately 30 sites in Japan. The patients should have received at least 1 cycle of chemotherapy and never receive immune oncology drug as 1st line treatment in stage IV. The patients will be enrolled continuously from the 1st patient who is enrolled in this study until target number of patients in each site.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20, Japanese men and women.
* Patients who have started at least 1 cycle of chemotherapy.
* Patients who provided informed consent by appropriate methods. In dead case, optout will be applicable.
* Patients who are diagnosed as stage IV (T4b, any N or any T, N2-3 or M1) UC between January 1st in 2017 and December 31st in 2018.
* Patients who have FFPE primary tumor sample collected after January 1st in 2017. The sample should be collected before any therapies including 1st line treatment in stage IV and therapies in stage III and other stages. It is possible to send sliced undyed section of primary tumor including 1 HE-stained section of same sample in case that patients cannot send FFPE primary tumor block.

Exclusion Criteria:

-Patients who are prior exposure to immune-mediated therapy as 1st line treatment in stage IV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a multi-center, non-interventional study, and Stage IV UC patients who have received at least 1 cycle of chemotherapy and have archived primary tumor sample collected after January 1st in 2017 will be of the interest. However, the patients who received immune oncology drug as 1st line treatment in stage IV will not be in this study.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Prevalence of PD-L1 in stage IV UC patients in real world setting. | Baseline
  Summarize number and calculate ratio of PD-L1 high or low/negative patients, respectively.

SECONDARY OUTCOMES:
Prevalence of TMB in stage IV UC patients in real world setting. | Baseline
  Calculate median and average of TMB levels. Summarize number and calculate ratio of TMB high or low/negative patients, respectively.
OS from start of 1st line treatment in stage IV | 2 years
  Median OS and OS rate at 12 months, 18 months and 24 months will be analysed based on Kaplan-Meier method and presented along with its 95% confidence interval.
PFS from start of 1st line treatment in stage IV | 18 months
  Median PFS and PFS rate at 6months, 12months and 18 months will be analysed based on Kaplan-Meier method and presented along with its 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Redacted Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419BR00014&attachmentIdentifier=193132e8-3b9c-4208-b0de-ab0b0f0b0e48&fileName=D419BR00014_YODO_redacted_synopsis.pdf&versionIdentifier=